CLINICAL TRIAL: NCT02960971
Title: DOLORISK: Understanding Risk Factors and Determinants for Neuropathic Pain - Neuropathic Pain After Lung Surgery
Brief Title: Neuropathic Pain After Lung Surgery
Status: Completed | Type: Observational
Sponsor: Danish Pain Research Center (Other)
Collaborators: DOLORisk Consortium (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DOLORISK-LUNG
Record Dates: First submitted 2016-11-08; First posted 2016-11-10 (Estimated); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Chronic Neuropathic Pain, Postoperative; Chronic Pain, Postoperative; Chronic Chemotherapy-induced Neuropathic Pain; Chronic Chemotherapy-induced Pain; Chronic Chemotherapy-induced Peripheral Neuropathy
MeSH Terms: conditions — Pain, Postoperative | interventions — Thoracic Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Thoracic surgery for lung cancer — Lung cancer resection performed via Video-assisted thoracoscopic surgery (VATS) and/or thoracotomy, including lobectomy, bilobectomy, pneumonectomy, resection of the tracheobronchial bifurcation, wedge resection, sleeve resection and combinations hereof.

SUMMARY:
To understand pain pathophysiology in terms of risk factors and protective mechanisms ranging from molecular pathways to societal impacts.

DETAILED DESCRIPTION:
Pain and loss of function are intimately associated with the reaction of the nervous system to neural damage. A lesion to the somatosensory nervous system caused by mechanical trauma, metabolic disease, neurotoxic chemicals, infection or tumor invasion may give rise to neuropathic pain. Neuropathic pain affects around 8% of the population and may negatively impact the individual's quality of life; moreover, the condition leads to significant costs to the healthcare system and society. Not all subjects with such a lesion develop neuropathic pain, and those who do develop neuropathic pain have varying degrees of symptom severity, impact and outcomes and may respond unpredictably to treatment.

The interaction between genetics and environmental and clinical factors in a susceptible individual most likely contribute to the variation in pain prevalence and severity. A better understanding of the exact nature of these risk factors and their interactions will ultimately improve the patients' health, both in terms of recognizing patients at risk and identifying new treatment modalities.

Genetic, neurophysiological and psychological factors all influence the risk of developing persistent pain. It is therefore possible to describe a genetic, neurophysiological and psychological profile, in particular in patients experiencing neuropathic pain after surgery and/or neurotoxic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects.
* Age ≥18 years.
* Patients scheduled for lung cancer resection performed via thoracoscopy and/or thoracotomy, including lobectomy, bilobectomy, pneumonectomy, resection of the tracheobronchial bifurcation, wedge resection, sleeve resection and combinations hereof.
* Willingness and ability to comply with study procedures as judged by the site investigator/manager.
* Expected availability for follow-up throughout the study, i.e., ~12 months.
* Willingness to voluntarily sign and date the study-specific informed consent form.

Exclusion Criteria:

* Mental incapacity or language barriers precluding adequate understanding of study procedures.
* Current alcohol or substance abuse according to the site investigator's medical judgement.
* Unsuitability for participation in the study for any other reason, e.g. due to a significant serious underlying condition (e.g. other cancer or AIDS), as determined by the site investigator/manager.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for lung cancer resection at the Department of Cardiothoracic and Vascular Surgery, Aarhus University Hospital, Denmark
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2021-06-16 (Actual)

PRIMARY OUTCOMES:
Chronic Neuropathic Pain, Postoperative | 12 months after surgery
  Neuropathic pain grading system, Finnerup et al. 2016 will be used.

SECONDARY OUTCOMES:
Chronic Chemotherapy-induced Peripheral Neuropathy | 12 months after surgery
  For case definition of neuropathy, Tesfaye et al. 2010 will be used.
Chronic Chemotherapy-induced Neuropathic Pain | 12 months after surgery
  Neuropathic pain grading system, Finnerup et al. 2016 will be used.
Acute Postoperative Pain | 0-5 days after surgery
  Rest and movement-evoked postoperative pain measured on an 11-point NRS
Area of peri-incisional hyperalgesia | 0-5 days after surgery
  Quantification of peri-incisional hyperalgesia - area and worst pin-prick pain intensity is assessed with a 5.88 monofilament

CONTACTS AND LOCATIONS:
Overall Officials: Nanna B Finnerup, DMSc, Study Director — Danish Pain Research Center, Aarhus University
Locations (2):
- Denmark (2):
  - Danish Pain Research Center, Aarhus University Hospital, Aarhus C
  - Department of Cardiothoracic and Vascular Surgery, Aarhus University Hospital, Aarhus N

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tesfaye S, Boulton AJ, Dyck PJ, Freeman R, Horowitz M, Kempler P, Lauria G, Malik RA, Spallone V, Vinik A, Bernardi L, Valensi P; Toronto Diabetic Neuropathy Expert Group. Diabetic neuropathies: update on definitions, diagnostic criteria, estimation of severity, and treatments. Diabetes Care. 2010 Oct;33(10):2285-93. doi: 10.2337/dc10-1303. PMID 20876709
- [Background] Finnerup NB, Haroutounian S, Kamerman P, Baron R, Bennett DLH, Bouhassira D, Cruccu G, Freeman R, Hansson P, Nurmikko T, Raja SN, Rice ASC, Serra J, Smith BH, Treede RD, Jensen TS. Neuropathic pain: an updated grading system for research and clinical practice. Pain. 2016 Aug;157(8):1599-1606. doi: 10.1097/j.pain.0000000000000492. PMID 27115670
- [Derived] Sperandio G, Baudic S, Bennedsgaard K, Grosen K, Andersen IS, Finnerup NB, Albi-Feldzer A, Flor H, Nees F, Bouhassira D, Attal N. Somatic and psychological predictors of chronic postsurgical pain in cancer patients: a machine learning approach in a longitudinal two-centre study. Br J Anaesth. 2026 Jan 7:S0007-0912(25)00847-5. doi: 10.1016/j.bja.2025.12.002. Online ahead of print. PMID 41506969
- See also: DOLORISK Consortium Homepage — http://www.dolorisk.eu